CLINICAL TRIAL: NCT06371612
Title: Comparison of the Effects of Ball Squeezing and Adhesive Remover Use on Pain and Fear in Children Aged 6-9 Years During the Removal of Peripheral Intravenous Cannula: A Randomised Experimental Study
Brief Title: Effects of Squeezing Ball and Using Adhesive Remover on Pain and Fear in Children Aged 6-9 Years During the Removal of Peripheral Intravenous Cannula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Guzide UGUCU, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MersinU*GUGUCU_004
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Procedural Pain; Fear of Pain
Keywords: pain; fear; children
MeSH Terms: conditions — Pain, Procedural; Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The children and their parents will be blinded to the groups. The principal researchers (R1, R2) will be blinded to the research hypotheses. The opaque envelopes are stored in a locked cabinet by the researcher who performed the randomization. Data entries will be performed using the codes A, B and C. Codes will be shared with the researchers after statistical analyses are conducted and the research report is written.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care (Active Comparator): First, the physical comfort of the children will be ensured in the invasive procedure room. In standard care practice, the parental presence is supported during all invasive procedures performed on children. Two minutes before the removal of the peripheral intravenous cannula, cotton balls soaked in antiseptic solution and squeezed will be gently applied to the fixation area.
  Interventions: Other: Standard Care
- Adhesive Remover Spray (Active Comparator): First, the physical comfort of the children will be ensured in the invasive procedure room. Two minutes prior to the removal of the peripheral intravenous cannula, an alcohol-free silicone-based aresol spray for medical use will be gently applied to the fixation site. The children will be supported by their parents.
  Interventions: Other: Adhesive Remover Spray
- Ball Squeezing + Adhesive Remover Spray (Experimental): : First, the physical comfort of the children will be ensured in the invasive procedure room. Two minutes prior to the removal of the peripheral intravenous cannula, an alcohol-free silicone-based aresol spray for medical use will be gently applied to the fixation site. At the same time, children will start squeezing the stress ball. The ball squeezing intervention will be terminated when the removal of the peripheral intravenous cannula is completed. The children will be supported by their parents.
  Interventions: Behavioral: Ball Squeezing + Adhesive Remover Spray

INTERVENTIONS:
Other: Standard Care — Parental Presence
  Arms: Standard Care
Other: Adhesive Remover Spray — Parental Presence + an alcohol-free silicone-based aresol spray for medical use
  Arms: Adhesive Remover Spray
Behavioral: Ball Squeezing + Adhesive Remover Spray — Parental Presence + an alcohol-free silicone-based aresol spray for medical use + squeezing the stress ball
  Arms: Ball Squeezing + Adhesive Remover Spray

SUMMARY:
Pediatric nurses have a key role in reducing pain related to interventions during the hospitalisation process. In this context, according to the type of invasive intervention, the nurse determines the appropriate non-pharmacological methods for the effective management of pain, taking into account the child's individuality, developmental stage and clinical presentation. For children during the hospitalisation process, the removal of a peripheral venous line is a painful and stressful experience, as is the insertion of a peripheral venous line. Children experience acute pain during the removal of hypoallergenic adhesives used for fixation of the peripheral venous line. The practice guideline recommends the use of alcohol-free silicone-based aerosol sprays for the removal of medical adhesive/ fixation materials (NICU Brain Sensitive Care Committee, 2015).

In this study, it was aimed to examine the effect of ball squeezing (active distraction) as a distraction method and the use of alcohol-free silicone-based aerosol adhesive remover spray on pain and fear in children aged 6-9 years during peripheral intravenous cannula removal.

DETAILED DESCRIPTION:
Research Hypotheses:

H1= There is a difference in the mean WB-FACES score during the procedure between the groups.

H2= There is a difference in the mean CFS score during the procedure between the groups.

Design and Settings: This parallel-group randomized trial will be conducted at the invasive procedure room of the pediatrics department of a university hospital. For this experimental research, 90 children aged 6-9 years will be assigned to three groups (Standard Care Group= SCG; n = 30, Adhesive Remover Spray Group = ARSG; n=30, and Ball Squeezing + Adhesive Remover Spray Group=BSG; n = 30) using block randomization.

Sample Size: The trial sample was calculated based on the study findings of "Ugucu, G., Uysal, D. A., Polat, O. G., Artuvan, Z., Kulcu, D. P., Aksu, D., ... & Temel, G. O. (2022). Effects of cartoon watching and bubble-blowing during venipuncture on pain, fear, and anxiety in children aged 6-8 years: a randomized experimental study. Journal of Pediatric Nursing, 65, e107-e114.". A priori power analysis was performed based on the effect size (d = 0.885, large effect) of the difference in pain scores between the groups (during the procedure). Using G*Power 3.1.9.7, the minimum sample size was calculated as 74 children, with 28 children per group, for a two-tailed hypothesis, an effect size of d = 0.885, an allocation ratio of n1/n2=1, type I error of 0.05, and a power of 90%. Considering that there may be drop-outs during the process, the number of groups was increased by 10%. The sample size of this study was determined as 90 children (30 children in each intervention group).

Data Collection Tools: It is decided to use the Child Information Form, Wong-Bakers FACES Pain Rating Scale and Child Fear Scale to collect the data. It includes "age, gender, previous experience of hospitalization, experience of procedural pain in last week, analgesic administration at least six hours before the procedure, size of peripheral IV needle, area of IV blood sample, parental presence during procedure, and baseline data of pain, anxiety and fear scores of children before procedure".

The Wong-Bakers FACES® Pain Rating Scale (WB-FACES): Developed by Wong and Baker in 1981 and revised in 1983, the instrument is used to assess physical pain in people who are communicative, responsive, and aged three years and older. The scale consists of faces ranging from "Face 0= no hurt" to "Face 10=hurts worst".

The Children's Fear Scale (CFS): The instrument assessed the pain-associated fear in children. Developed by McMurty et al. (2011), the Turkish validity-reliability study of this visual scale was conducted by Özalp-Gerçeker et al. (2018) and it is scored from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome.

Interventions: The invasive procedure room in the clinic which decorated with cartoon characters and ornaments on the walls will be used. The intervention can be administered to only one child at a time in the room. In routine practice, the parental presence is supported during all invasive procedures performed on children. However, the nurses' uniforms have a print/pattern of cartoon characters in the routine practice. The room will have the same characteristics for all children and their parents in terms of environmental conditions such as light, temperature, noise, and seat. Before the procedure, children's pain, and fear will be assessed after providing developmentally appropriate information. The parents will be also informed about how to support their children. The same researchers will be performed the removal of peripheral intravenous cannula (R1) and observational pain and fear assessments (R2) in all children. R1 and R2 are nurses with more than five years of experience in pediatrics and degrees in scientific fields (MScN, PhD).

Standard Care Group: First, the physical comfort of the children will be ensured in the invasive procedure room. In standard care practice, the parental presence is supported during all invasive procedures performed on children. Two minutes before the removal of the peripheral intravenous cannula, cotton balls soaked in antiseptic solution and squeezed will be gently applied to the fixation area.

Adhesive Remover Spray Group: First, the physical comfort of the children will be ensured in the invasive procedure room. Two minutes prior to the removal of the peripheral intravenous cannula, an alcohol-free silicone-based aresol spray for medical use will be gently applied to the fixation site. The children will be supported by their parents.

Ball Squeezing + Adhesive Remover Spray Group: First, the physical comfort of the children will be ensured in the invasive procedure room. Two minutes prior to the removal of the peripheral intravenous cannula, an alcohol-free silicone-based aresol spray for medical use will be gently applied to the fixation site. At the same time, children will start squeezing the stress ball. The ball squeezing intervention will be terminated when the removal of the peripheral intravenous cannula is completed. The children will be supported by their parents.

Ethical Considerations: The study was granted approval by the ethics committee and written institutional permission by the hospital. Parents and children will be informed about the procedure and that they could withdraw from the study at any time without explanation. Written consent of parents and verbal consent of children before the study will be obtained.

Statistical Methods: The statistical significance level was determined as 0.05. Kolmogrow-Smirnov test will be used in the normality analysis of dependent variables. Chi-square and comparison of means tests will be used to determine the similarity of the groups. Appropriate parametric or non-parametric tests will be used according to the normality of the distribution in the comparison of means between groups and within groups. In case of differences in the averages between groups, the effect size appropriate to the test family will be used.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6-9 years
* Child with need or plan for the removal of the peripheral intravenous cannula (antecubital fossa of arm, superficial dorsal venous of hand)

Exclusion Criteria:

* Child with a neurodegenerative disease, mental retardation, vision and hearing problems, chronic, life-threatening (sepsis, shock, respiratory / cardiac arrest) or genetic disease
* Child with use of opioids, narcotics, analgesics or sedatives in the last 24 hours before the procedure

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | during the removal of the peripheral intravenous cannula
  The Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Fear by Children's Fear Scale | during the removal of the peripheral intravenous cannula
  The Child Fear Scale was used.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to 4 (extreme fear). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Pain assesed by Wong-Baker FACES | at 2nd minutes after the removal of the peripheral intravenous cannula
  The Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Fear by Children's Fear Scale | at 2nd minutes after the removal of the peripheral intravenous cannula
  The Child Fear Scale was used.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to 4 (extreme fear). Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Guzide UGUCU, PhD, MScN, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Guzel Polat O, Ugucu G, Akdeniz Uysal D, Polat N, Tuzun O, Sonmez Duzkaya D, Celebioglu A. Effects of using an adhesive remover spray and squeezing a stress ball on pain and fear of pain during peripheral intravenous cannula removal in children aged 6-9 years: A randomized controlled trial. J Pediatr Nurs. 2025 Sep-Oct;84:23-29. doi: 10.1016/j.pedn.2025.05.009. Epub 2025 May 16. PMID 40381428